CLINICAL TRIAL: NCT02296307
Title: Diagnosing Ovarian & Endometrial Cancer Early (DOvEE) by Targeting Symptomatic Women
Brief Title: DOvEE - Diagnosing Ovarian & Endometrial Cancer Early
Acronym: DOvEE
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Lucy Gilbert, Professor, Department of Obstetrics and Gynecology, McGill University
Other Study IDs: CIHR-276061
Record Dates: First submitted 2014-10-28; First posted 2014-11-20 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Neoplasms
Keywords: Aged; Algorithms; CA-125 Antigen/blood*; Chi-Square Distribution; Early Detection of Cancer*; Feasibility Studies; Female; Humans; Logistic Models; Mass Screening/methods*; Middle Aged; Neoplasm Grading; Neoplasm Invasiveness; Neoplasm Staging; Ovarian Neoplasms/diagnosis*; Ovarian Neoplasms/epidemiology; Ovarian Neoplasms/immunology; Ovarian Neoplasms/ultrasonography; Pilot Projects; Predictive Value of Tests; Prevalence; Prognosis; Prospective Studies; Quebec/epidemiology; Tumor Burden
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Invasiveness; Disease | interventions — CA-125 Antigen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DOvEE Participants: All symptomatic women who are eligible for participation in the DOvEE trial receive the same interventions:
  Blood test: CA-125 biomarker at day 1 and week 6-8. Second Test: Transvaginal Ultrasound at day 1. Follow-up Phone Call: Confirms continuing health 6 months after last visit.
  Interventions: Other: Blood test: CA-125 biomarker; Other: Second Test: Transvaginal Ultrasound; Other: Follow-up phone call

INTERVENTIONS:
Other: Blood test: CA-125 biomarker — * CA-125 biomarker blood test at visit 1, day 1.
  * CA-125 biomarker blood test at visit 2, week 6.
  Other Names: CA125; CA 125; cancer antigen 125; carbohydrate antigen 125
Other: Second Test: Transvaginal Ultrasound — -Transvaginal Ultrasound at visit 1, day 1.
Other: Follow-up phone call — Phone call 6 months after last visit to verify continued health.

SUMMARY:
This study hopes to improve early detection of ovarian and endometrial cancers. It will determine if women with bloating, abdominal distension, abdominal/pelvic pain, increased urinary frequency and/or early satiety, benefit from earlier surgery after screening by CA-125 ovarian cancer biomarker and transvaginal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an approved informed consent form (ICF).
2. Be ≥ 45 years of age.
3. Have at least one symptom outlined in below for a period of ≥2 weeks but ≤ 1 year:

   * Feeling full after eating only a few bites, loss of appetite
   * Diarrhea, constipation, bowel or rectum feels full, change in bowel habits, constant urge to have a bowel movement, painful or burning bowel movements, rectal pain, painful defecation
   * Bloating, distension of abdomen, clothes around the waist feel too tight, feel an abdominal mass
   * Weight loss not because of dieting
   * Nausea, vomiting, heartburn, gas, burping, indigestion
   * Increased urinary frequency, need to urinate urgently, pressure on the bladder, leaking urine, burning sensation when urinating, need to urinate but unable to do so, unable to empty bladder completely, feeling full after urinating
   * Vaginal discharge, bleeding, spotting, deep pain on intercourse
   * Discomfort or pain in abdomen, or pelvic region, or lower back
4. Subjects must be willing to comply with study protocol

Exclusion Criteria:

1. Previous bilateral salpingo-oophorectomy (BSO)
2. Previous diagnosis of cancer in the ovaries, fallopian tubes, or peritoneum
3. Current bleeding per rectum, not due to haemorrhoids
4. Current frank haematuria
5. Symptoms that suggest the need for urgent clinical evaluation outside of a research protocol

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are 45+ years of age, living in greater Montreal. Women may self-identify and contact the DOvEE Study directly, or be referred from primary care or physicians or specialists.
Sampling Method: Non-Probability Sample
Enrollment: 13600 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of diagnoses in early, curable stage. | Up to 3 years
  To determine whether the provision of fast-track diagnostic evaluation of symptomatic women ≥50 years will result in a higher proportion of ovarian cancer, including high-grade serous cancers (HGSCs), diagnosed in low-volume, completely resectable stage.

SECONDARY OUTCOMES:
Number of participants with physical morbidity related to the program as a measure of safety and tolerability | Up to 6 weeks
  To determine the physical morbidity associated with testing symptomatic women for ovarian cancer by CA-125 and transvaginal ultrasound.
  Participants will complete the DOvE Program Impact Assessment at Visit 1, and the Impact of Program on Patient's Well-being Questionnaire at Visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Gilbert, MD,MSc,FRCOG, Principal Investigator — McGill University
Locations (8):
- Canada (8):
  - West Island Cancer Wellness Centre, Kirkland, Quebec
  - Axion 50 plus, Laval, Quebec
  - Clinique Familiale Pas-A-Pas, Montreal, Quebec
  - Clinique Médicale du Haut-Anjou, Montreal, Quebec
  - McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec
  - Queen Elizabeth Health Centre, Montreal, Quebec
  - Lachine Hospital, Montreal, Quebec
  - Clinique du Dr. L. Quintal, Saint-Lambert, Quebec

REFERENCES:
- [Background] Gilbert L, Basso O, Sampalis J, Karp I, Martins C, Feng J, Piedimonte S, Quintal L, Ramanakumar AV, Takefman J, Grigorie MS, Artho G, Krishnamurthy S; DOvE Study Group. Assessment of symptomatic women for early diagnosis of ovarian cancer: results from the prospective DOvE pilot project. Lancet Oncol. 2012 Mar;13(3):285-91. doi: 10.1016/S1470-2045(11)70333-3. Epub 2012 Jan 17. PMID 22257524